CLINICAL TRIAL: NCT06025422
Title: Evaluation of Footwear Fit Guidelines Under Pressure in At-Risk Feet
Brief Title: In-shoe Pressures Associated With Footwear Fit Guidelines
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Salford (Other)
Responsible Party: Sponsor
Other Study IDs: edge136945; 20/0006190 (Other Grant/Funding Number: Diabetes UK); 273255 (Other: Health Research Authority (IRAS no.))
Record Dates: First submitted 2023-05-11; First posted 2023-09-06 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer; Diabetic Neuropathies
Keywords: in-shoe peak plantar pressure; plantar thermal stress response; diabetes footwear fit; toe gap
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
One in five foot ulcers are caused by the footwear worn by people with diabetes, yet there is a lack of consensus around footwear fit. Recommended toe gaps (the gap between the longest toe and the inside of the shoe) vary depending on the footwear guidance referred to but no research to date has assessed the recommendations' effectiveness in minimising in-shoe pressures.

The investigators will carry out a pilot study in 60 people with diabetes and loss of foot sensation (neuropathy). In this study, the investigators will measure in-shoe pressures whilst participants walk at the same pace to the beat of a metronome. An insole placed inside participants' shoes will measure in-shoe pressures. Participants will wear the same (standardised) type of footwear. The study is designed to detect a difference in pressure within this made-to-measure footwear whose fit conforms to Standard 1 guidance compared with footwear whose fit conforms to Standard 2 guidance. Differences between Standards 1 and 2 with Standard 3 will be considered secondary analyses. Standards are simplified to three non-overlapping recommended toe gap ranges of 0.5-1.0cm; 1.5-2.0cm and 1.0-1.5cm.

The investigators will also analyse the heat images taken with a thermographic camera before and after walking in standardised footwear whose fit confirms to these standards (this is known as the plantar thermal stress response to walking). Footwear fit will be determined by measuring the dimensions of participants' feet and that of participants' footwear and comparing the two.

The investigators will also measure footwear fit and associated in-shoe pressure/plantar thermal stress response in participants' habitual footwear during walking at paced and self-selected speeds.

DETAILED DESCRIPTION:
The investigators will recruit 60 participants with diabetes, neuropathy and a history of ulceration. The investigators will set a minimum target recruitment number for each sex (25 minimum for each).

People with diabetes and neuropathy will be recruited through the Leicester General Hospital Multi-disciplinary Foot Team (MDFT). Leicestershire Partnership NHS Trust (LPT) will be used as a PIC site which runs 24 Community Podiatry clinics to identify possible participants. Our CODEC database (an ongoing trial looking at the effect of sleep patterns on blood glucose control) where participants agreed to be contacted regarding other studies will also be used to identify possible participants.

Participants who consent to participate in the study, will have foot measurements. These foot measurements taken at baseline are both relevant to footwear fit and necessary to order comfortable, custom fit standardised house shoes aimed at those with diabetes who are at risk. Those participants assigned to footwear fit Standards which are within the IWGDF recommended range of 1.0-2.0cm toe gap will also be permitted to retain their made-to-measure standardised footwear - a house shoe designed for people with diabetes with at-risk feet. Participants assigned footwear with a non-IWGDF compliant footwear fit (i.e. a short toe gap of less than 1.0cm) will not be permitted to retain their standardised footwear given uncertainty regarding their suitability for long-term use.

The air-conditioning will be switched on to control the ambient temperature. Participants will be asked to bring everyday (i.e. most frequently used) footwear or prescribed footwear.

Participants' habitual footwear will then be photographed by a member of the research team using a CE-marked digital camera and the footwear style, condition and materials are recorded by a researcher using the Footwear Assessment Form (FAF). Footwear fit will then be determined by measuring the internal length of the shoe using a special gauge and measuring internal shoe width using a calliper-type device. Heel height will also be measured using a ruler.

Carbon impression sheets will be used to measure foot posture by capturing the outline of the foot. The participant will be asked to remove any socks with assistance to help with this if necessary.

A special insole that measures pressure will be slipped into the participant's footwear.The participant will walk within habitual footwear at normal everyday walking pace and paced using a metronome at a specific normal walking pace. In-shoe pressures will be monitored and recorded throughout.

The participant will then walk whilst wearing standardised footwear (identical for all participants) again with metronome pacing. The participant will then complete a few questionnaires to say how comfortable and easy to use both the trainers and habitual footwear are. The participant will be asked to stand upon a carbon sheet which captures an impression of feet whilst standing in a relaxed posture.

Thermal images of participants' feet are taken after ten minutes of acclimatization.

Participants will don the thin, seamless cotton socks provided. The pressure monitoring insoles are then placed in the participant's habitual footwear. The participant will be asked to complete 4 walks at a self-selected pace during which in-shoe pressures are measured. The participant will then be asked to walk some additional steps until reaching a total of 200 steps. A thermal image is then taken of the feet immediately after removal of both habitual footwear and socks.

Participants are then asked to repeat this process, except this time the participant is paced by the sound of a metronome to walk at a pre-selected pace. On completion, a thermal image is again taken of participants' feet immediately after removal of habitual footwear and socks.

Participants will be asked to rate the comfort of habitually worn footwear by completing a survey. A member of the research team will be on hand to answer any questions participants may have regarding the survey. Participants will rate habitually worn footwear using usability and comfort surveys. As before, a member of the research team will be available to answer any questions regarding the survey.

After putting on the thin, seamless cotton socks provided, pressure monitoring insoles are then placed in the standardised footwear provided for the participant. Participants will now be asked to put on standardised footwear and assisted if necessary. Participants will be given some time to acclimatize to the new footwear. The participant will be asked to rate the comfort of the standardised footwear using the Comfort Survey before beginning the walking trial. Assuming there are no problems, the walking trial will proceed.

The participant will once again walk to the beat of the metronome for a total of 200 steps (split into 4 trials capturing midgait steps, plus additional steps). On completion, a thermal image is again taken of their feet immediately after they have removed both habitually worn footwear and socks. If a participant has trouble with the pacing, the investigators may ask the participant to walk more additional trials but these will not exceed the total of 200 steps. After a short foot check, participants will then put any socks and habitually worn footwear back on. Participants will rate standardised footwear using the usability survey. As before, a member of the research team will be available to answer any questions regarding the survey. This completes participants' tasks in the study.

Where in-shoe pressures within study participants' habitual footwear are found to be in excess of 200 kPa threshold associated with an increased risk of ulceration, the investigators will refer the participant to the Podiatry Service enclosing an in-shoe pressure image depicting the location of the highest pressure regions to assist in devising offloading measures such as therapeutic insoles and orthotics. This referral does not form part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-80 years
* Confirmed diagnosis of diabetes mellitus type 1 or type 2
* Confirmed diagnosis of neuropathy;
* Able to walk unaided for a minimum of 200 steps with capacity to attend the research site
* PAR-Q physical activity questionnaire does not indicate any possible heart problems, dizziness or other issue indicating unsuitability for mild physical exercise involved in walking
* Willingness and capacity to participate in the study and to sign the informed consent form

Exclusion Criteria:

* Unconfirmed diabetes mellitus diagnosis
* Inability to ambulate independently without walking aids
* Presence of rheumatoid arthritis
* Active ulcer (i.e. having an active ulcer at the time of recruitment)
* Recently healed ulcer (an ulcer which has had less than six months to fully heal)
* History of Charcot in foot/joints
* Previous minor or major amputation
* Neurological disorders other than diabetes-related neuropathy potentially affecting gait, balance or posture
* Evidence of significant peripheral vascular disease e.g. (i) attendance at a specialist vascular clinic; (ii) documentation of occlusive arterial disease or intervention; (iii) at least one pulse should be palpable on the affected foot with exclusion where neither pulse is palpable
* Blood pressure >180/100 or <90/50
* Unable to understand written and verbal English
* PAR-Q physical activity questionnaire indicates possible heart problems, dizziness or other issue indicating unsuitability for mild physical exercise involved in walking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty people with diabetes type 1 or 2 and neuropathy aged between 18 and 80
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
During the procedure difference in mean in-shoe PPP associated with each toe gap standard within standardised footwear @ regulated pace | During the procedure, peak plantar pressure in kilopascals (kPa) is measured with Novel Pedar pressure measuring insoles and software whilst completing 4 x 12 midgait steps at a speed of 2 miles per hour +/- 5%
  During the procedure Difference in the mean average in-shoe peak plantar pressure (PPP) associated with each toe gap standard (measured by Pedar-X pressure monitoring insoles) during walking within standardised footwear at a regulated pace
During the procedure difference in the mean in-shoe PPP by ROI associated with each toe gap standard | During the procedure, peak plantar pressure in kilopascals (kPa) is measured with Novel Pedar pressure measuring insoles and software whilst completing 4 x 12 midgait steps at a speed of 2 miles per hour +/- 5%
  During the procedure Mean in-shoe peak plantar pressure (PPP) for each region of interest (ROI) (comprising 10 regions: hallux, toes 2/3, toes 4/5, metatarsal 1, metatarsal 2/3, metatarsal 4/5, medial midfoot, lateral midfoot, medial heel, lateral heel) associated with each toe gap standard during walking within standardised footwear at a regulated pace

SECONDARY OUTCOMES:
During the procedure Exploratory secondary analysis of toe gap Standard 3 in relation to toe gap Standards 1 and 2 | During the procedure, peak plantar pressure in kilopascals (kPa) is measured with Novel Pedar pressure measuring insoles and software whilst completing 4 x 12 midgait steps at a speed of 2 miles per hour +/- 5%
  During the procedure Differences in mean average in-shoe peak plantar pressure associated with toe gap Standards 1 and 2 with Standard 3 will be considered secondary analyses.
During the procedure Pressure time integral & contact area associated with toe gap standards in standardised footwear | During the procedure, peak plantar pressure in kilopascals (kPa) is measured with Novel Pedar pressure measuring insoles and software whilst completing 4 x 12 midgait steps at a speed of 2 miles per hour +/- 5%
  During the procedure Pressure time integral and contact area associated with each toe gap standard during walking within standardised footwear at a regulated pace
During the procedure Proportion of participants with in-shoe PPP > 200 kilopascals in standardised footwear | During the procedure, peak plantar pressure in kilopascals (kPa) is measured with Novel Pedar pressure measuring insoles and software whilst completing 4 x 12 midgait steps at a speed of 2 miles per hour +/- 5%
  During the procedure The proportion of participants where the mean in-shoe peak plantar pressure (PPP) at the forefoot, toes or metatarsal regions exceeds 200 kPa or for the plantar region as a whole during walking in standardised footwear at a regulated pace
During the procedure PTSR associated with each toe gap standard in standardised footwear | Thermal image taken with FLIR T540-EST thermal camera of plantar surface of feet at rest and after 200 steps within standardised footwear
  During the procedure Plantar thermal stress response (PTSR) is defined as changes in 95th percentile temperature values in Celsius when comparing thermal images of the plantar surface of the feet at rest prior to walking and a thermal image of the feet after walking for each region of interest (forefoot, midfoot, rearfoot) associated with each toe gap standard whist walking in standardised footwear at regulated pace
During the procedure Mean in-shoe PPP within habitual footwear at a self-selected and regulated pace | During the procedure, peak plantar pressure in kilopascals (kPa) is measured with Novel Pedar pressure measuring insoles and software whilst completing 4 x 12 midgait steps at a speed of 2 miles per hour +/- 5%
  During the procedure Mean in-shoe peak plantar pressure overall and for each region of interest (comprising 10 regions: hallux, toes 2/3, toes 4/5, metatarsal 1, metatarsal 2/3, metatarsal 4/5, medial midfoot, lateral midfoot, medial heel, lateral heel) associated with each toe gap standard during walking within habitual footwear at a self-selected and regulated pace
During the procedure Proportion of participants with in-shoe PPP > 200 kilopascals in habitual footwear | During the procedure, peak plantar pressure in kilopascals (kPa) is measured with Novel Pedar pressure measuring insoles and software whilst completing 4 x 12 midgait steps at a speed of 2 miles per hour +/- 5%
  During the procedure The proportion of participants where the mean in-shoe peak plantar pressure at the forefoot, toes or metatarsal regions exceeds 200 kPa or for the plantar region as a whole during walking in habitual footwear at a regulated and self-selected pace
During the procedure Pressure time integral & contact area associated with toe gap standards in habitual footwear | During the procedure, pressure time integral and contact area is measured with Novel Pedar pressure measuring insoles and software whilst completing 4 x 12 midgait steps at a speed of 2 miles per hour +/- 5%
  During the procedure Pressure time integral and contact area associated with each toe gap standard during walking within habitual footwear at a regulated pace
During the procedure Percentage of participants with incorrectly fitted / correctly fitted habitual footwear | At presentation on visit 2
  During the procedure The percentage of participants with incorrectly fitted / correctly fitted habitual footwear as defined by each standard and the mean, minimum, maximum and standard deviation of toe gaps found within their habitual footwear
During the procedure PTSR associated with habitual footwear | Thermal image taken with FLIR T540-EST thermal camera of plantar surface of feet at rest and after 200 steps within habitual footwear
  During the procedure Plantar thermal stress response (PTSR) is defined as changes in 95th percentile temperature values in Celsius when comparing thermal images of the plantar surface of the feet at rest prior to walking and a thermal image of the feet after walking for each region of interest (forefoot, midfoot, rearfoot) associated with each toe gap standard whist walking in habitual footwear

CONTACTS AND LOCATIONS:
Overall Officials: Petra J Jones, Principal Investigator — University Hospitals, Leicester
Locations (1):
- Leicester Diabetes Centre, Leicester, Leicestershire, United Kingdom